CLINICAL TRIAL: NCT06937372
Title: Delivery and Implementation of a Randomised Cluster Crossover Trial on Thrombosis
Brief Title: Delivery and Implementation of a Randomised Crossover Trial on Thrombosis
Acronym: DIRECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Edge Number: 177790; NIHR159321 (Other Grant/Funding Number: NIHR Health Technology Assessment (HTA) Programme)
Record Dates: First submitted 2025-04-10; First posted 2025-04-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hip Fractures; Venous Thromboembolism (VTE)
Keywords: Hip fracture; Blood clot; Aspirin; Low molecular weight heparin (LMWH)
MeSH Terms: conditions — Hip Fractures; Venous Thromboembolism; Thrombosis | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: A multicentre, pragmatic, standard-of-care controlled, cluster (hospital) randomised, single crossover, registry-enabled trial reporting a single-sided comparison for non-inferiority of a first-line thromboprophylaxis strategy including aspirin compared with LMWH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin Arm (Experimental): Patients in hospitals allocated to this arm will receive aspirin as their routine thromboprophylaxis after surgery. Aspirin is a widely available, low-cost medication that may reduce the risk of blood clots with fewer side effects such as bleeding.
  Interventions: Drug: Patients in hospitals allocated to this arm will receive aspirin as their routine thromboprophylaxis after surgery.
- Low Molecular Weight Heparin (LMWH) Arm (Active Comparator): Patients in hospitals allocated to this arm will receive LMWH, which is the current standard treatment in many hospitals for preventing blood clots after hip surgery.
  Interventions: Drug: Low molecular weight heparin (LMWH)

INTERVENTIONS:
Drug: Patients in hospitals allocated to this arm will receive aspirin as their routine thromboprophylaxis after surgery. — Unlike low molecular weight heparin (LMWH), which requires daily subcutaneous injections, aspirin is taken orally, making it more comfortable and acceptable for patients, particularly the elderly or those with mobility issues. Aspirin is significantly less expensive than injectable anticoagulants like LMWH or newer oral anticoagulants, making it a potentially cost-effective alternative for thromboprophylaxis.
  Arms: Aspirin Arm
Drug: Low molecular weight heparin (LMWH) — LMWH is administered via daily subcutaneous injection, typically starting shortly after surgery and continued for a defined period as per each hospital's local policy, often 14 to 28 days. LMWH has a proven track record of reducing the risk of deep vein thrombosis (DVT) and pulmonary embolism (PE) after surgery.
  However, it carries a risk of bleeding and may be challenging for some frail or elderly patients to tolerate, especially if self-injection is required post-discharge.
  Arms: Low Molecular Weight Heparin (LMWH) Arm

SUMMARY:
What is the Study About? The DIRECT study (Delivery and Implementation of a Randomised Crossover Trial on Thrombosis) is a large research project investigating the best way to prevent blood clots (thrombosis) in people who break their hip. The study will compare two common treatments: aspirin (a tablet) and low molecular weight heparin (LMWH, an injection).

Every year, thousands of people in the UK suffer a hip fracture, which often requires surgery and hospital care. After a hip fracture, patients are at risk of developing serious blood clots in their legs (deep vein thrombosis, DVT) or lungs (pulmonary embolism, PE), which can be life-threatening. Currently, doctors prescribe different medications to prevent these clots, but there is uncertainty about which treatment is best for people with hip fractures.

Why is This Study Needed? Blood clot prevention is vital for hip fracture patients, but the current recommended treatment (LMWH) involves daily injections for 28 days, which some patients find uncomfortable and difficult to manage at home. Aspirin, a tablet taken by mouth, is a much simpler alternative, but there is not enough evidence to confirm whether it is as effective and safe as LMWH in this group of patients.

The DIRECT study will help doctors and the NHS understand whether aspirin could be a safe and cost-effective alternative to LMWH. If aspirin is found to be just as effective, it could make treatment easier for patients and save millions of pounds for the NHS.

How Will the Study Work? The study will involve 96 hospitals across the UK and will include over 21,000 patients aged 60 and older who have broken their hip. Hospitals will be randomly assigned to use either aspirin or LMWH as their standard treatment for a set period. After this, they will switch to the other treatment. This approach allows researchers to compare the two treatments fairly.

All data will be collected from national NHS databases, which routinely record patient care and outcomes. This means patients will not need to do anything extra or attend additional follow-ups.

What Are the Expected Benefits?

This study will provide clear evidence on which treatment is better for preventing blood clots while minimising risks like bleeding. If aspirin is shown to be as effective as LMWH, it could:

* Reduce the need for daily injections, making treatment more comfortable for patients.
* Lower NHS costs, as aspirin is much cheaper than LMWH.
* Provide a simple, widely available treatment option for older adults with hip fractures.

How Will Patient Data Be Protected? The study will use anonymised patient data from NHS records. This means that all personal details will be kept confidential and protected according to strict NHS and research regulations. Patients who do not want their data to be used can opt out via NHS data-sharing policies.

Summary The DIRECT study is an important project that will help improve care for hip fracture patients by determining whether aspirin can be a safe and effective alternative to injections for preventing blood clots. The results will help shape future NHS guidelines, ensuring patients receive the best possible treatment while reducing unnecessary costs and discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 60 to 150 years sustaining fragility hip fracture identified by their entry into UK hip registries.

Exclusion Criteria:

* Individuals who do not meet the eligibility criteria to be enrolled in the NHFD and SHFA registries Hip fracture individuals above 150 years of age.

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21194 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary Composite Outcome: 90-Day Symptomatic Venous Thromboembolism (VTE) and All-Cause Mortality | 28 days (safety) and 90 days (efficacy)
  To estimate and draw inferences on the risk differences between first-line venous thromboembolism (VTE) thromboprophylaxis management strategies including aspirin versus low molecular weight heparin (LMWH) of the co-primary outcomes of VTE events, combined pulmonary embolism (PE) and deep vein thrombosis (DVT), within 90 days (efficacy) and major bleeding events within 28 days (safety) after hospital admission following index hip fracture.

SECONDARY OUTCOMES:
Cause-Specific Mortality | 90 days
  Deaths specifically attributable to pulmonary embolism, bleeding, or other identifiable causes within 90 days post-surgery
Major Bleeding Events | 28 days
  Incidents of clinically significant bleeding requiring medical intervention or transfusion.